CLINICAL TRIAL: NCT03467477
Title: A Multicenter Screening Study With Flortaucipir F 18 in Patients With Early Symptomatic AD; #2
Brief Title: Tau Screening Study in Subjects With Early Symptomatic AD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18F-AV-1451-A24
Record Dates: First submitted 2018-03-08; First posted 2018-03-16 (Actual); Results first posted 2020-08-24 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Flortaucipir PET Scan (Experimental)
  Interventions: Drug: Flortaucipir F18; Procedure: Brain PET Scan

INTERVENTIONS:
Drug: Flortaucipir F18 — 370 megabecquerel (MBq) IV single-dose
  Other Names: 18F-AV-1451; [F-18]T807; LY3191748
Procedure: Brain PET Scan — positron emission tomography (PET) scan of the brain

SUMMARY:
This protocol is designed to serve as a pre-screening study for subjects who are potentially eligible for Alzheimer's Disease (AD) therapeutic trials that require tau imaging for inclusion by means of a flortaucipir F18 Positron Emission Tomography (PET) scan.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with gradual and progressive change in memory function reported by the patient or informant for ≥6 months
2. Patients who have a mini-mental status exam (MMSE) score between 20-28 inclusive
3. Patients who are willing to undergo a PET scan using flortaucipir F 18
4. Patients who give informed consent or have a legally authorized representative (LAR) available to consent at the time of enrollment
5. A study partner who must be available if the patient enters the treatment trial

Exclusion Criteria:

1. Are females of childbearing potential who are not surgically sterile, not refraining from sexual activity or not using reliable methods of contraception. Females of childbearing potential must not be pregnant (negative serum β-HCG [beta human chorionic gonadotropin] at screening and negative urine β-HCG prior to flortaucipir F 18 injection) or breastfeeding at screening. Females should agree to avoid becoming pregnant by refraining from sexual activity or using reliable contraceptive methods for 24 hours following administration of flortaucipir F 18 injection;
2. Patients who lack, in the investigator's opinion, adequate premorbid literacy, adequate vision, or adequate hearing to complete the required psychometric testing;
3. Have significant neurological disease affecting the central nervous system (CNS), other than AD, that may affect cognition or ability to complete the study, including but not limited to, other dementias, serious infection of the brain, Parkinson's disease, multiple concussions, or epilepsy or recurrent seizures (except febrile childhood seizures);
4. Patients with any current primary psychiatric diagnosis other than AD if, in the judgment of the investigator, the psychiatric disorder or symptom is likely to confound interpretation of drug effect, affect cognitive assessment, or affect the patient's ability to complete the study [Patients with history of schizophrenia or other chronic psychosis are excluded.];
5. Have a current serious or unstable illness including, cardiovascular, hepatic, renal, gastroenterologic, respiratory, endocrinologic, neurologic (other than AD), psychiatric, immunologic, or hematologic disease and other conditions that, in the investigator's opinion, could interfere with the analyses in this study; or has a life expectancy of <24 months;
6. Has a history of cancer within the last 5 years, with the exception of nonmetastatic basal and/or squamous cell carcinoma of the skin, in situ cervical cancer, non-progressive prostate cancer, or other cancers with low risk of recurrence or spread;
7. Have a past history (suspected or confirmed) of Hepatitis B or Hepatitis C;
8. Are clinically judged by the investigator to be at serious risk for suicide as assessed by medical history, examination, or the Columbia-Suicide Severity Rating Scale (C-SSRS).
9. Have a history of alcohol or drug disorder (except tobacco use disorder) within 2 years before the screening visit;
10. Have a history of clinically significant multiple or severe drug allergies or severe post treatment hypersensitivity reactions (including but not limited to erythema multiforme major, linear immunoglobulin A dermatosis, toxic epidermal necrolysis, and/or exfoliative dermatitis)
11. Have known positive serologic findings for human immunodeficiency virus (HIV) antibodies. Local laws and regulations may apply to whether testing is required.
12. Has previous MRI evidence of significant abnormality that would suggest another potential etiology for progressive dementia or a clinically significant finding that may impact the patient's ability to safely participate in the study;
13. Have any contraindications for MRI, including claustrophobia or the presence of contraindicated metal (ferromagnetic) implants/cardiac pacemaker;
14. Have any clinically important abnormality at screening, as determined by investigator, in physical or neurological examination, vital signs, ECG, or clinical laboratory test results that could be detrimental to the patient, could compromise the study, or show evidence of other etiologies for dementia.
15. Has hypersensitivity to flortaucipir F 18 or any of its excipients;
16. Intend to use drugs known to significantly prolong the QT interval within 14 days or 5 half-lives, whichever is longer, of a scheduled screening/baseline flortaucipir F 18 PET scan, or have medical history of risk factors for torsades de pointes.
17. Have an ECG corrected QT (QTcF) interval measurement >450 msec (men) or >470 msec (women) at screening (as determined at the investigational site).
18. Have poor venous access;
19. Contraindication to PET;
20. Present or planned exposure to ionizing radiation that, in combination with the planned administration of study PET ligands, would result in a cumulative exposure that exceeds local recommended exposure limits;
21. Patients that are currently enrolled in any other interventional clinical trial involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study
22. Have participated, within the last 30 days in a clinical trial involving an investigational product. If the previous investigational product is scientifically or medically incompatible with this study and has a long half-life, 3 months or 5 half-lives (whichever is longer) should have passed prior to screening (Participation in observational studies may be permitted upon review of the observational study protocol and approval by the sponsor).
23. Are investigator site personnel directly affiliated with this study and/or their immediate families; immediate family is defined as spouse, parent, child, or sibling whether biological or legally adopted;
24. Are Lilly employees or are employees of third-party organizations (TPOs) involved in a study that requires exclusion of their employees;
25. In the opinion of the investigator, are otherwise unsuitable for a study of this type.
26. Have received treatment with a stable dose of an acetylcholinesterase inhibitor (AChEI) and/or memantine for less than 1 months [If a patient has recently stopped an AChEI and/or memantine, he or she must have discontinued treatment at least 1 months prior].
27. Have changes in concomitant medications that could potentially affect cognition and their dosing should be stable for at least 1 month before screening, (does not apply to medications with limited duration of use, such as antibiotics).
28. Have received active immunization agents for the treatment of Alzheimer's Disease
29. Have known allergies to LY3303560, related compounds, or any components of the formulation; or history of significant atopy
30. Have allergies to either monoclonal antibodies, diphenhydramine, epinephrine, or methylprednisolone;
31. Are receiving Immunoglobulin G therapy (also known as gamma globulin or intravenous immunoglobulin [IVIG])

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Chair — Avid Radiopharmaceuticals
Locations (9):
- United States (9):
  - Irvine Center for Clinical Research, Irvine, California
  - Brain Matters Research, Delray Beach, Florida
  - Neuropsychiatric Research Center of Southwest Florida, Fort Myers, Florida
  - Renstar Medical Research, Ocala, Florida
  - BioClinica Research, Orlando, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Cotton O'neil Clinical Research Center, Topeka, Kansas
  - Butler Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment occurred between Mar 2018 and Nov 2018. Recruited subjects with clinically diagnosed early AD who were interested in participating in AD therapeutic clinical trials being conducted by Eli Lilly and Company.
Groups:
- Early Symptomatic AD Subjects: Early Symptomatic AD subjects in the flortaucipir PET scan arm
Period: Overall Study
Arm/Group | Early Symptomatic AD Subjects
Started | 161
Completed | 161
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Early Symptomatic AD Subjects
Number analyzed (Participants) | 161
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.0 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93
  Male | 68
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 154
  More than one race | 0
  Unknown or Not Reported | 0
MMSE [Mean (Standard Deviation); unit: units on a scale] — Mini-mental status exam (MMSE) is a 30-point questionnaire that is used to measure cognitive impairment. Scores range from 0 to 30 with lower scores representing greater levels of cognitive impairment.
  units on a scale | 25.0 (2.51)

OUTCOME MEASURES:

1. Primary Outcome: Flortaucipir Qualitative Results (Visual Reads)
Description: Flortaucipir PET scans were rated visually by an expert reader as follows: Not consistent with an AD pattern (τAD-), Moderate AD pattern (τAD+), or Advanced AD pattern and likely to progress (τAD++). Eligibility for future studies was determined from the flortaucipir PET scan according to protocol-specified criteria.
Time Frame: baseline scan
Measure: Count of Participants; unit: Participants
Groups:
- Early Symptomatic AD, Eligible for Future Trials: Subjects determined to be eligible for future studies from the flortaucipir PET scan arm.
- Early Symptomatic AD, Ineligible for Future Trials: Subjects who were not eligible for future studies from the flortaucipir PET scan arm.
- Early Symptomatic AD, Not Evaluable: Subjects determined to be not eligible for future studies from the flortaucipir PET scan arm due to unevaluable PET scan for quantitation
- Early Symptomatic AD (Total): All subjects with early symptomatic AD from the flortaucipir PET scan arm
Arm/Group | Early Symptomatic AD, Eligible for Future Trials | Early Symptomatic AD, Ineligible for Future Trials | Early Symptomatic AD, Not Evaluable | Early Symptomatic AD (Total)
Number analyzed (Participants) | 55 | 105 | 1 | 161
Participants
  τAD++, advanced AD pattern | 51 | 13 | 1 | 65
  τAD+, moderate AD pattern | 4 | 10 | 0 | 14
  τAD-, pattern not consistent with AD | 0 | 82 | 0 | 82

2. Primary Outcome: Flortaucipir Quantitative Results (SUVr)
Description: Flortaucipir standardized uptake value ratio (SUVr). A value of 1 signifies no flortaucipir activity above background, values greater than 1 signify increasing flortaucipir activity in the brain. Visual read categories as described for previous measure.
Time Frame: baseline scan
Population: SUVr was not collected for patients with a τAD- result (n=82) and one subject had an unevaluable flortaucipir scan for quantitation. Therefore, analysis population n=78.
Measure: Mean (Standard Deviation); unit: standardized uptake value ratio (SUVr)
Arm/Group | Early Symptomatic AD, Eligible for Future Trials | Early Symptomatic AD, Ineligible for Future Trials | Early Symptomatic AD, Not Evaluable | Early Symptomatic AD (Total)
Number analyzed (Participants) | 55 | 23 | 1 | 78
standardized uptake value ratio (SUVr)
  SUVr all subjects: number analyzed (Participants) | 55 | 23 | 0 | 78
  SUVr all subjects | 1.24766 (0.122786) | 1.38020 (0.343791) |  | 1.28674 (0.219185)
  SUVr τAD++ subjects: number analyzed (Participants) | 51 | 13 | 0 | 64
  SUVr τAD++ subjects | 1.25687 (0.122501) | 1.64935 (0.187100) |  | 1.33659 (0.209539)
  SUVr τAD+ subjects: number analyzed (Participants) | 4 | 10 | 0 | 14
  SUVr τAD+ subjects | 1.13025 (0.038043) | 1.03031 (0.039727) |  | 1.05886 (0.060181)

ADVERSE EVENTS:
Time Frame: 48 hours after study drug administration
Description: Adverse events (AEs) were collected at scan visits, regardless of attribution to study drug. End of study for AE reporting was 48 hours after the last study drug administration. AEs occurring after study drug administration, but outside that window were not recorded, unless considered attributable to study drug.
Groups:
- Safety Analysis Population: All subjects with early symptomatic AD from the flortaucipir PET scan arm who received one dose of flortaucipir
Arm/Group | Safety Analysis Population
All-Cause Mortality (participants affected / at risk) | 0/161
Serious Adverse Events (participants affected / at risk) | 0/161
Other Adverse Events (participants affected / at risk) | 2/161
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Analysis Population (N=161)
claustrophobia (Psychiatric disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/77/NCT03467477/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-11): https://cdn.clinicaltrials.gov/large-docs/77/NCT03467477/SAP_001.pdf